CLINICAL TRIAL: NCT00869544
Title: Pneumocystis in Pathogenesis of HIV-associated Emphysema
Acronym: PACT
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Alison Morris, Professor, University of Pittsburgh
Other Study IDs: IRB0606151; 5R01HL083461-05 (NIH)
Record Dates: First submitted 2009-03-25; First posted 2009-03-26 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: HIV Infections; Pneumocystis Pneumonia; Emphysema; Chronic Obstructive Pulmonary Disease; Asthma
Keywords: HIV; smoker; emphysema; antiretrovirals; COPD
MeSH Terms: conditions — HIV Infections; Pneumonia, Pneumocystis; Emphysema; Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — oral wash blood sputum BAL
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- HIV: Those positive for HIV and those negative but at high risk for HIV. Both positive and negative for HIV who smoke and those who do not smoke. Both HIV positive and negative with and without asthma and/or COPD

SUMMARY:
A. Statement of Hypotheses:

HIV-infected patients have an increased incidence of emphysema compared to non-HIV-infected smokers, and it has been hypothesized that this accelerated disease progression is the result of one or more latent infections that amplifies the pulmonary inflammatory response to cigarette smoke. Pneumocystis is one infectious agent that likely plays a key role in the development of HIV-associated emphysema. Colonization with Pneumocystis has been demonstrated in HIV-infected subjects, and HIV-infected smokers are particularly susceptible to Pc colonization regardless of CD4 cell count or use of prophylaxis. Pneumocystis colonization is also increased in non-HIV-infected patients with chronic obstructive pulmonary disease (COPD) and is directly related to the severity of the disease. The presence of Pneumocystis in the lungs, even at low levels as seen in colonization, produces inflammatory changes similar to those seen in COPD, with increases in the numbers of neutrophils and cytotoxic CD8+ lymphocytes. We propose that Pneumocystis accelerates emphysema in HIV-infected smokers by stimulating inflammation and tissue destruction. We will examine the role of co-infection with Pneumocystis in the pathogenesis of HIV-associated emphysema and the mechanism by which it causes emphysema progression. These studies will lead to information that will provide a rational basis for prevention and therapy of HIV-associated emphysema and provide a model for emphysema in the general population

DETAILED DESCRIPTION:
We propose that Pneumocystis accelerates emphysema in HIV-infected smokers by stimulating inflammation and tissue destruction. This grant will examine the role of co-infection with Pneumocystis in the pathogenesis of HIV-associated emphysema and the mechanism by which it causes emphysema progression. These studies will lead to information that will provide a rational basis for prevention and therapy of HIV-associated emphysema and provide a model for emphysema in the general population

antiretroviral therapy (HAART), impressive declines in morbidity and mortality from HIV have been seen [18]. These improvements do not constitute a cure, however; and over 400,000 people are currently living with HIV in the United States and there are 40 million people infected worldwide. With improved treatment and increases in life expectancy, incidence of other types of lung diseases such as HIV-associated emphysema and pulmonary hypertension may become more common. Respiratory symptoms are extremely common in the HIV-infected population, even among those without a history of pulmonary infections. HIV-infected subjects have been noted to have an accelerated form of chronic obstructive pulmonary disease (COPD)/emphysema [4, 5]. This disease is seen in those with untreated HIV disease and may become more common in the treated HIV population as it has frequently been reported in those without a history of AIDS-related pulmonary complications.

Smoking-related diseases such as emphysema are of particular concern in the HIV+ population. Smoking rates are high in this population and long term exposure to cigarette smoke in the setting of HIV infection may increase the number of complications seen. Smoking in the HIV+ population is associated with worse general health, physical functioning, quality of life, and cognitive functioning Before the HAART era, HIV+ subjects were noted to have an accelerated form of emphysema. Unlike many of the AIDS-defining opportunistic infections, HIV-associated emphysema may actually be more common in the current era of HIV as it is frequently reported in those without a history of AIDS-related pulmonary complications and because the aging HIV+ population has a longer exposure to smoking and HIV. HIV-associated emphysema was identified as a critical area for future research by a recent NIH workshop on pulmonary complications of HIV.

Whether emphysema continues to be increased in the HIV+ population in the HAART era is unknown. We hypothesize that emphysema may actually have increased as subjects live longer with chronic pulmonary exposure to the virus, to smoking, and to the inflammation that occurs in even treated HIV+ patients. We believe that prevalence will be increased compared to HIV- controls and that progression will be accelerated. Assessment of degree of emphysema and its distribution can be accomplished using quantitative CT morphometry density analysis. This technique measures lung density by pixel analysis expressed in Hounsfield units (HU) or its inverse (ml of gas/gram of tissue) which increases proportionately with the magnitude of emphysema. These measurements have been histologically-verified and give quantitative, reproducible measurements of percentage and distribution of lung considered normal, mildly emphysematous, and severely emphysematous. By adding the lung images to this protocol, we will be maximizing the information gained from this study with minimal increases in risk or subject inconvenience.

Pneumocystis jirovecii Based on our preliminary data in humans and primates, we believe that Pneumocystis (Pc) is one infectious agent that is critical in the pathogenesis of HIV-associated emphysema. Pneumocystis jirovecii (formerly known as Pneumocystis carinii f. sp. hominis)[19] is a eukaryotic pathogen that causes pneumonia in immunocompromised hosts. Despite the fact that PCP is responsible for a large degree of morbidity and mortality in immunosuppressed populations, little is understood about the organism's epidemiology. The recent development of molecular techniques to identify and genotype Pc has provided an important tool with which to explore the epidemiology of the organism. Polymerase chain reaction (PCR) detects low numbers of organisms, particularly in cases where routine histochemical staining methods are negative [21, 22]. Use of PCR, particularly nested PCR, for detection of Pc has led to discovery of the organism among asymptomatic subjects. The rate of colonization in asymptomatic HIV-infected subjects appears to be higher than that seen in the general population with estimates ranging from 12 to 46% depending on the subject population and respiratory samples studied [11, 12, 14, 16, 22].

Evidence linking HIV-associated emphysema and Pc colonization Pathogenesis of HIV-associated emphysema is not understood. The disease is likely multifactorial with contributions from smoking, HIV infection, and subclinical infections. Based on several lines of preliminary data, we believe that Pc plays a key role in development of HIV-associated emphysema. The evidence linking Pc and emphysema includes the high rates of both emphysema and Pc colonization in HIV-infected smokers, COPD-like changes that occur after PCP, an increase in Pc colonization in COPD that corresponds to disease severity and is independent of smoking history, and similarity between the inflammatory response in Pc colonization and COPD. The role of Pc colonization in HIV-associated emphysema has not been tested directly.

With the completion of the human genome project and advances in human genetic research, it is now possible for us to conduct comprehensive population genetic studies aimed at the identification of genetic factors associated with development of, and outcomes from, different diseases. Separately, newer technologies such as Luminex, microarray, SAGE, and proteomic analyses have made it possible to study expression profiles of thousands of genes. Simultaneous development of statistical methods to detect patterns of gene expression and link these patterns with clinical outcomes, have facilitated the identification of prognostic markers of disease (e.g. breast cancer and BRCA-1, and markers of tumor metastasis in melanoma). In particular, these studies both elucidate the mechanisms of disease pathogenesis, as well as identify targets for potential therapeutic intervention. It is crucial to the success of these scientific endeavors to link the cellular, protein, and gene expression and genetic data to clinical and demographic data on a large substrate of subjects, or the interpretation and results of these statistical analyses will be flawed.

ELIGIBILITY:
Inclusion Criteria:

* Subject is Male / Female 18years of age or older.
* Subject has been previously determined to be HIV-infected or has been participating in the Pitt Men's study or is seen at the UPMC HIV/AIDS program

Exclusion Criteria:

* Subject is experiencing acute onset of shortness of breath, cough, fevers or heart conditions problems such as tachycardia, angina or arrhythmias
* Female subject has told us she is pregnant (this might affect pulmonary function values,we will not require pregnancy testing.)
* Subject has had an MI, CVA, or cardiovascular event within the past 3 months.
* Subject has had eye or abdominal surgery within past 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who have been determined to attend the UPMC HIV/AIDS program and/or participants in the Pitt Mens study.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2007-08; Primary Completion 2010-09 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Pc colonization | 5 years
  The main endpoints that will be assessed are the extent of Pc colonization in this population and its relationship to lung function, inflammatory cells and cytokines, and proteases.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Morris-Gimbel, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Montefiore Hospital, CTRC MUH, Keystone Bldg., Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Gingo MR, Lucht L, Daly KR, Djawe K, Palella FJ, Abraham AG, Bream JH, Witt MD, Kingsley LA, Norris KA, Walzer PD, Morris A. Serologic responses to pneumocystis proteins in HIV patients with and without Pneumocystis jirovecii pneumonia. J Acquir Immune Defic Syndr. 2011 Jul 1;57(3):190-6. doi: 10.1097/QAI.0b013e3182167516. PMID 21372726
- [Background] Morris A, Netravali M, Kling HM, Shipley T, Ross T, Sciurba FC, Norris KA. Relationship of pneumocystis antibody response to severity of chronic obstructive pulmonary disease. Clin Infect Dis. 2008 Oct 1;47(7):e64-8. doi: 10.1086/591701. PMID 18724825
- [Background] Morris A, Gingo MR, George MP, Lucht L, Kessinger C, Singh V, Hillenbrand M, Busch M, McMahon D, Norris KA, Champion HC, Gladwin MT, Zhang Y, Steele C, Sciurba FC. Cardiopulmonary function in individuals with HIV infection in the antiretroviral therapy era. AIDS. 2012 Mar 27;26(6):731-40. doi: 10.1097/QAD.0b013e32835099ae. PMID 22210636
- [Background] Gingo MR, Wenzel SE, Steele C, Kessinger CJ, Lucht L, Lawther T, Busch M, Hillenbrand ME, Weinman R, Slivka WA, McMahon DK, Zhang Y, Sciurba FC, Morris A. Asthma diagnosis and airway bronchodilator response in HIV-infected patients. J Allergy Clin Immunol. 2012 Mar;129(3):708-714.e8. doi: 10.1016/j.jaci.2011.11.015. Epub 2011 Dec 15. PMID 22177327
- [Derived] Gingo MR, Nouraie M, Kessinger CJ, Greenblatt RM, Huang L, Kleerup EC, Kingsley L, McMahon DK, Morris A. Decreased Lung Function and All-Cause Mortality in HIV-infected Individuals. Ann Am Thorac Soc. 2018 Feb;15(2):192-199. doi: 10.1513/AnnalsATS.201606-492OC. PMID 29313714